CLINICAL TRIAL: NCT05600387
Title: Empagliflozin on the Function of Left Atrium in Heart Failure With Mildly Reduced or Preserved Ejection Fraction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Zhijun Sun (Other)
Responsible Party: Sponsor-Investigator, Zhijun Sun, Director of the second Department of cardiovascular medicine, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022PS1015K
Record Dates: First submitted 2022-10-21; First posted 2022-10-31 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure; Heart Failure With Preserved Ejection Fraction; Heart Failure With Mid Range Ejection Fraction
Keywords: Heart Failure; Empagliflozin; Function of left atrium
MeSH Terms: conditions — Heart Failure | interventions — empagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin group (Experimental): subjects in Empagliflozin group take 10mg Empagliflozin 10mg per day
  Interventions: Drug: Empagliflozin 10 MG
- Control group (No Intervention): subjects in Control group will not receive Empagliflozin or other sglt-2 inhibitors

INTERVENTIONS:
Drug: Empagliflozin 10 MG — subjects in Empagliflozin group take 10mg Empagliflozin per day
  Arms: Empagliflozin group

SUMMARY:
The number of heart failure with mildly reduced or preserved ejection fraction gradually increases. SGLT2-i has been shown to reduce the risk of hospitalization for heart failure and cardiovascular death among patients with chronic heart failure and a left ventricular ejection fraction of 40% or more . However,its effect on the function on left atrium in heart failure with mildly reduced or preserved ejection fraction is still unknown.

DETAILED DESCRIPTION:
Heart failure with mildly reduced or preserved ejection fraction has become an important part of heart failure, the proportion is also gradually increased .Atrial fibrillation , as a common arrhythmia disease, is often caused by heart failure and aggravates the process of heart failure. It has been documented that in patients with heart failure and an ejection fraction more than 40%, it may have a higher incidence of atrial fibrillation.Heart failure and atrial fibrillation together increase the risk of stroke, hospitalization for heart failure, and all-cause death from heart failure.

SGLT-2 inhibitor (SGLT-2i) is a new metabolic drug, through a variety of mechanisms on cardiac metabolism, has been shown to reduce the risk of death and rehospitalization, and improve the health of patients with heart failure.But the effect on preventing arrhythmia in patients with heart failure is still unclear. Some studies have shown that SGLT-2i reduces the left atrial volume index and the left ventricular diastolic volume index compared with placebo and some have proved that the indicators of the function of left atrium, such as peak atrial longitudinal strain (PALS), peak atrial contraction strain (PACS), can effectively predict the occurrence of atrial fibrillation. The purpose of this study is to apply empagliflozin (a class of SGLT-2i) in heart failure patients with mildly reduced or preserved ejection fraction to measure the changes in the function of left atrium and thus verify its prevention and control effect on atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, BMI18.5-27.9kg/m²
* Meet the definition of chronic heart failure and an ejection fraction of 40% or more (according to 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure)
* Elevated NT-proBNP levels of more than 300 pg/mL
* Signed and dated written informed consent form

Exclusion Criteria:

* Myocardial infarction,coronary artery bypass graft surgery, or other major cardiovascular surgery within 30 days after enrollment
* Percutaneous coronary intervention ,coronary artery bypass graft surgery,cardiac resynchronization therapy, implantable cardioverter defibrillatoror or other cardiac surgeries within 90 days prior to enrollment
* Atrial fibrillation or flutter
* SGLT-2i using within 90 days prior to enrollment
* Cardiomyopathy based on infiltrative diseases (e.g. amyloidosis), accumulation diseases (e.g. haemochromatosis, Fabry disease),cardiomyopathy with reversible causes (e.g. stress cardiomyopathy), or known pericardial constriction
* Acute decompensated heart failure.
* Moderate to severe valvular stenosis or regurgitation
* Symptomatic hypotension with systolic pressure ≤ 90mmHg or uncontrolled hypertension using drugs with systolic blood pressure of ≥180 mmHg at randomization
* Sever infectious diseases(e.g. Severe myocarditis, severe pneumonia, and severe urinary tract infection)
* Chronic pulmonary disease requiring home oxygen, oral corticosteroid therapy or hospitalization for exacerbation within 12 months
* Other significant co-morbid conditions(impaired renal function( an estimated glomerular filtration rate of <20 mL/min/1.73 m2), hepatic failure, malignant tumors, severe hematologic diseases, etc.)
* Major surgery performed within 90 days prior to enrollment or major scheduled elective surgery within 90 days after enrollment(major according to the investigator's assessment,such as gastrointestinal surgery that might interfere with trial medication absorption or malignant tumors surgery)
* Type 1 diabetes or history of ketoacidosis
* Pregnancy
* Completion within 90 days of a trial of another drug study. Receipt of any investigative treatment other than the study medications for this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-05 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
change of peak atrial longitudinal strain during 6 months | 6 months
  peak atrial longitudinal strain will be assessed using echocardiography
change of peak atrial contraction strain during 6 months | 6 months
  peak atrial contraction strain will be assessed using echocardiography
change of left atrial conduit strain during 6 months | 6 months
  left atrial conduit strain will be assessed using echocardiography

SECONDARY OUTCOMES:
change of left atrial volume index during 6 months | 6 months
  left atrial volume index will be assessed using echocardiography
change of E/A during 6 months | 6 months
  E/A will be assessed using echocardiography，and it is defined as the ratio of peak early diastolic flow velocity and peak late diastolic flow velocity
change of E/e'during 6 months | 6 months
  E/e' will be assessed using echocardiography and it is defined as the ratio of peak early diastolic flow velocity and peak early diastolic mitral annular velocity
change of left ventricular global longitudinal strain during 6 months | 6 months
  left ventricular global longitudinal strain will be assessed using echocardiography
change of left ventricular ejection fraction during 6 months | 6 months
  left ventricular ejection fraction will be assessed using echocardiography
peak atrial longitudinal strain in the sixth month | 6 months
  peak atrial longitudinal strain will be assessed using echocardiography
peak atrial contraction strain in the sixth month | 6 months
  peak atrial contraction strain will be assessed using echocardiography
left atrial conduit strain in the sixth month | 6 months
  left atrial conduit strain will be assessed using echocardiography
left atrial volume index in the sixth month | 6 months
  left atrial volume index will be assessed using echocardiography
E/A in the sixth month | 6 months
  E/A will be assessed using echocardiography，and it is defined as the ratio of peak early diastolic flow velocity and peak late diastolic flow velocity
E/e' in the sixth month | 6 months
  E/e' will be assessed using echocardiography and it is defined as the ratio of peak early diastolic flow velocity and peak early diastolic mitral annular velocity
left ventricular global longitudinal strain in the sixth month | 6 months
  left ventricular global longitudinal strain will be assessed using echocardiography
left ventricular ejection fraction in the sixth month | 6 months
  left ventricular ejection fraction will be assessed using echocardiography
new-onset atrial fibrillation in the sixth month | 6 months
  new-onset atrial fibrillation is defined as follows:no atrial fibrillation at screening and electrocardiogram in the sixth month indicates atrial fibrillation

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No